CLINICAL TRIAL: NCT06518759
Title: Effect of Glossopharyngeal Versus Diaphragmatic Breathing Exercise on Pulmonary Function After Decortication Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mai Gamal El-Din Mostafa, Principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/003896
Record Dates: First submitted 2024-07-17; First posted 2024-07-24 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2024-07

CONDITIONS: Pulmonary Disease
MeSH Terms: conditions — Lung Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Traditional chest techniques (Active Comparator): the patients will receive traditional chest techniques only
  Interventions: Other: traditional chest techniques
- Traditional chest techniques +Glossopharyngeal breathing exercise (Experimental): the patients will receive traditional chest techniques and glossopharyngeal breathing exercise
  Interventions: Other: traditional chest techniques; Other: Glossopharyngeal breathing exercise
- Traditional chest techniques +diaphragmatic breathing exercise (Experimental): the patients will receive traditional chest techniques and diaphragmatic breathing exercise
  Interventions: Other: traditional chest techniques; Other: Diaphragmatic breathing exercise

INTERVENTIONS:
Other: traditional chest techniques — patients will receive traditional chest techniques in the form of percussion and vibration, 2 times per day, 3 sets 5 repetitions per each set for 20 minutes, 3 times per week for 2 weeks
Other: Glossopharyngeal breathing exercise — patients will receive Glossopharyngeal breathing exercise, 2 times per day, 3 sets 5 repetitions per each set for 20 minutes, 3 times per week for 2 weeks.
  Arms: Traditional chest techniques +Glossopharyngeal breathing exercise
Other: Diaphragmatic breathing exercise — patients will receive diaphragmatic breathing exercise, 2 times per day, 3 sets 5 repetitions per each set for 20 minutes, 3 times per week for 2 weeks.
  Arms: Traditional chest techniques +diaphragmatic breathing exercise

SUMMARY:
This study will be conducted to compare between the effect of glossopharyngeal and diaphragmatic breathing exercises on pulmonary functions after decortication surgery

DETAILED DESCRIPTION:
Lung decortication is a well-known procedure for the treatment of empyema. Persistent lung collapse and non-expansion of the lung parenchyma are frequently noticed in the postoperative period after decortications, chest physiotherapy plays a crucial role in the re-expansion of underlying parenchyma.

There is an increased flow of patients after decortication surgery to hospitals who suffer from decreased lung volumes so the hospitalization period for them increases which puts an economical burden on health insurance services with a decreased level of quality of life that is the most concern to improve patient status and relieve this burden. So this study aims to improve patient's lung volumes and arterial blood gas parameters which improves patient status through two various forms of breathing exercises.

ELIGIBILITY:
Inclusion Criteria:

* The participant's body mass index (BMI) will be ranged from 25- 29.9 kg/m2
* The patient will receive treatment after 24 hours after decortication
* The study will be in the intensive care unit (ICU).
* The patients have unilateral lung decortication
* Their vital capacity is 70% or less.

Exclusion Criteria:

* Cancerous patient.
* Inability to comprehend and follow instructions as in dementia
* paralytic involvement of thorax muscle
* Abdominal diseases that affect diaphragmatic function
* Diaphragmatic paralysis

Ages: 40 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2024-07-30 (Actual); Primary Completion 2025-03-15 (Actual); Study Completion 2025-03-31 (Actual)

PRIMARY OUTCOMES:
Tidal volume | within 2 weeks
  The spirometer device (Meditech, made in China) will be used to measure tidal volume for all participants in all groups before and after the treatment program. It is the amount of air that moves in or out of the lungs with each respiratory cycle. It measures about 400 ml in a healthy female.
Inspiratory reserve volume (IRV) | within 2 weeks
  The spirometer device (Meditech, made in China) will be used to measure inspiratory reserve volume (IRV) for all participants in all groups before and after the treatment program.
  - IRV: It is the amount of air that can be forcibly inhaled after normal tidal volume. The normal adult value is 1900-3300 ml.
Expiratory reserve volume (ERV) | within 2 weeks
  The spirometer device (Meditech, made in China) will be used to measure expiratory reserve volume (ERV) for all participants in all groups before and after the treatment program.
  ERV: It is the amount of extra air above normal breath-exhaled during forceful breath out, its average is about 800ml in females.
Measurement of the potential of hydrogen (PH) | within 2 weeks
  Blood gas analyzer will be used to measure the potential of hydrogen (PH) for all participants in all groups before and after the treatment program.
  The blood sample was taken from the radial or brachial or femoral artery or from arterial catheter and put in the device.
  The normative value of pH is7.35-7.45
Measurement of the partial arterial pressure of carbon dioxide(PaCO2) | within 2 weeks
  Blood gas analyzer will be used to measure the partial arterial pressure of carbon dioxide(PaCO2) for all participants in all groups before and after the treatment program.
  The blood sample was taken from the radial or brachial or femoral artery or from arterial catheter and put in the device.
  the normative value of PaCO2 is 4.7-6 KPa.
Measurement of the partial arterial pressure of oxygen (PaO2) | within 2 weeks
  Blood gas analyzer will be used to measure the partial arterial pressure of oxygen (PaO2)for all participants in all groups before and after the treatment program.
  The blood sample was taken from the radial or brachial or femoral artery or from arterial catheter and put in the device.
  the normative value of Pao2 is 1.7-13.3 KPa.
Measurement of the Bicarbonate (HCO3) | within 2 weeks
  Blood gas analyzer will be used to measure the Bicarbonate (HCO3) for all participants in all groups before and after the treatment program.
  The blood sample was taken from the radial or brachial or femoral artery or from arterial catheter and put in the device.
  The normative value of HCO3 is 22-26 mmol/L.
Measurement of oxygen saturation (SO2) | within 2 weeks
  Blood gas analyzer will be used to measure oxygen saturation (SO2) for all participants in all groups before and after the treatment program.
  The blood sample was taken from the radial or brachial or femoral artery or from arterial catheter and put in the device.
  The normative value of SO2 is 95-100%..

CONTACTS AND LOCATIONS:
Overall Officials: Nesreen El-Nahas, professor, Study Chair — Cairo University
Locations (1):
- Mai Gamal El-Din Mostafa, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol